CLINICAL TRIAL: NCT03997149
Title: Stress-induced Eating Behavior: Implications for Pediatric Obesity Disparities
Brief Title: Stress Reactivity Study in Adolescents
Acronym: SRAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rebecca Hasson, Director, Childhood Disparities Research Laboratory, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HUM00078153
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Stress; Eating Behavior
Keywords: Trier Social Stress Test
MeSH Terms: conditions — Feeding Behavior | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: Participants completed a stress condition and rest condition in random order.
Who Masked: Participant
Masking Description: Immediately following each condition, participants were provided with snacks to eat at their leisure. Participants were not told that their post-condition food consumption would be measured and was part of the research study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Condition (Experimental): The stress condition involved the Trier Social Stress Test (TSST), a standardized laboratory stressor designed to elicit psychological stress and cortisol responses. Following the TSST, participants were brought to a separate room, instructed to rest and given the option to eat at their leisure. Books and magazines were included in the room for the participant to utilize.
  Interventions: Behavioral: Acute Laboratory Stressor
- Rest Condition (Placebo Comparator): Participants completed a control condition on a separate day. This condition followed the same sequence of events as the stress condition with the exception that the 20-minute TSST was replaced with a 20-minute low-affect educational film screening.
  Interventions: Behavioral: Low affect video

INTERVENTIONS:
Behavioral: Acute Laboratory Stressor — The TSST was 20 minutes long and consisted of a five-minute instructional period where participants listened to a pre-recorded tape; a five-minute speech preparation period; a five-minute challenging serial subtraction task; and a five-minute videotaped public speaking task in front of a panel of three evaluative, non-affirming judges dressed in white coats.
  Other Names: Trier Social Stress Test
  Arms: Stress Condition
Behavioral: Low affect video — The 20-minute TSST was replaced with a 20-minute low-affect educational film screening.
  Arms: Rest Condition

SUMMARY:
The goal of this study was to examine the glucocorticoid and behavioral responses to a psychological stressor in obese African-American and non-Latino white adolescents. Participants were exposed to the Trier Social Stress Test (TSST) and a control condition on separate days. Immediately following each condition, participants were provided with snacks to eat at their leisure. Reactivity was assessed via salivary cortisol and alpha-amylase area under the curve (AUC), and adolescents were categorized as high or low reactors.

DETAILED DESCRIPTION:
In the United States, pediatric obesity has more than tripled in the last 30 years, particularly among certain racial/ethnic groups including African-Americans. This disparity is partially attributable to greater exposure to psychological stress reported in this group (relative to non-Latino whites). Chronic psychological stress leads to weight gain directly through prolonged exposure to biological stress mediators such as cortisol and indirectly through behavioral pathways involving cortisol-induced increases in food consumption. An exciting arena of scientific advancements is focusing on identifying the specific pathways through which chronic stress influences eating behavior with emerging evidence to suggest that food intake, which is commonly increased during periods of stress, may serve as one key mechanism linking stress and obesity, particularly in African-American youth who are disproportionately exposed to chronic stress and have greater access to, and consumption of, energy-dense palatable foods. It is critical to advance understanding of the interplay between stress and food intake in understanding racial/ethnic disparities in pediatric obesity because stress eating represents a modifiable health behavior. That is, increased food intake during periods of elevated stress can be targeted for intervention in ways that may ameliorate the deleterious effects of stress on obesity risk. This project investigated the role of stress eating as a pathway linking chronic stress and obesity in African-American and non-Latino white adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese adolescents ages 14- 19 years

Exclusion Criteria:

* Currently pregnant
* Had been enrolled in a weight loss program in the last 6 months
* Were current smokers (e.g., tobacco, marijuana, vaping)
* Were diagnosed with a mental health condition (e.g, depression)
* Were diagnosed with a chronic condition known to affect weight, appetite, blood glucose or insulin levels (e.g., diabetes)
* Were taking medications known to affect metabolic processes (e.g., growth hormone, ritalin, metformin, etc)
* Had food allergies, intolerances, or other dietary restrictions

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Food consumption | 2 hours
  Change in grams of each food consumed during the control and stress conditions were recorded and calories were calculated using the corresponding nutritional labels.

SECONDARY OUTCOMES:
Salivary cortisol area under the curve | 2 hours
  During the control and stress conditions, saliva samples were taken at times 10, 25, 58, 88 and 118 minutes after arrival to analyze cortisol responses to the TSST. Area under the curve was calculated from the initial cortisol sample collected to the final cortisol sample collected: [AUC=(x2+x1)/(t2-t1) + (x3+x2)/(t3-t2) + (xk+xj)/(tk-tj)].
Salivary alpha amylase area under the curve | 2 hours
  During the control and stress conditions, saliva samples were taken at times 10, 25, 58, 88 and 118 minutes after arrival to analyze alpha amylase responses to the TSST. Area under the curve was calculated from the initial alpha-amylase sample collected to the final alpha amylase sample collected [AUC=(x2+x1)/(t2-t1) + (x3+x2)/(t3-t2) + (xk+xj)/(tk-tj)].

OTHER OUTCOMES:
Heart rate area under the curve | 2 hours
  Heart rate was taken throughout the control and stress conditions. Area under the curve was calculated from the initial heart rate collected to the final heart rate sample collected [AUC=(x2+x1)/(t2-t1) + (x3+x2)/(t3-t2) + (xk+xj)/(tk-tj)].
Blood pressure area under the curve | 2 hours
  Blood pressure was taken throughout the control and stress conditions. Area under the curve was calculated from the initial blood pressure reading collected to the final blood pressure reading collected [AUC=(x2+x1)/(t2-t1) + (x3+x2)/(t3-t2) + (xk+xj)/(tk-tj)].

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hasson, PhD, Principal Investigator — University of Michigan
Locations (1):
- Childhood Disparities Research Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified participant data will be shared with other researchers during data analysis and manuscript preparation.